CLINICAL TRIAL: NCT04716062
Title: Short-term and Oncological Outcomes of Laparoscopic Colorectal Cancer Surgery in Obese Patients
Acronym: Surg_2021
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliera Specializzata in Gastroenterologia Saverio de Bellis (Other)
Responsible Party: Principal Investigator, Gianluigi Giannelli, Medical Doctor, Professor, Azienda Ospedaliera Specializzata in Gastroenterologia Saverio de Bellis
Other Study IDs: Surg_2021
Record Dates: First submitted 2021-01-14; First posted 2021-01-20 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Obesity; Colorectal Cancer
MeSH Terms: conditions — Obesity; Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- subjects who underwent open-air surgery: Fifty-one (37%) out of 138 subjects underwent open-air surgery.
  Interventions: Procedure: Open or Laparoscopic-assisted Colorectal surgery
- subjects underwent laparoscopic-assisted surgery: A total of 87 (63%) out of 138 subjects underwent laparoscopic-assisted surgery.
  Interventions: Procedure: Open or Laparoscopic-assisted Colorectal surgery

INTERVENTIONS:
Procedure: Open or Laparoscopic-assisted Colorectal surgery — Colorectal surgery

SUMMARY:
A total of 138 consecutive patients who underwent laparoscopic-assisted or open colectomy for colorectal cancer (CRC) were included in the present study. Subjects commonly shared a condition of overweight or obesity. The investigators aimed to define any difference between the two different groups (open vs laparoscopic-assisted surgery) and a series of outcomes, i.e. hospitalization, Lymph nodes number, Intra-Surgery complications, and Clavien Dindo score.

DETAILED DESCRIPTION:
A total of 138 consecutive patients who underwent laparoscopic-assisted or open colectomy for colorectal cancer (CRC) were included in the present study. Intra-Surgery complications, Previous surgery, Readmission Post Intervention, Location of surgery, Duration of Surgery, Re-intervention (yes), Clearance, and CRM were collected. Subjects commonly shared overweight or obesity. The investigators aimed to define any difference between the two different groups (open vs laparoscopic-assisted surgery) and a series of outcomes, i.e. hospitalization, Lymph nodes number, Intra-Surgery complications, and Clavien Dindo score.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index >25 Kg/m2
* Colorectal cancer (CRC)

Exclusion Criteria:

* Current emergency conditions (i.e., perforation and\or occlusion)
* Pregnancy,
* Co-existing peritoneal carcinomatosis
* Contraindications to LS, such as cardiorespiratory comorbidities (CHD, CHF, and other severe CVD)
* Prior transverse resections

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 138 overweight or obese subjects. Fifty-one (37%) subjects underwent open-air surgery and 87 (63%) to VL surgery.
Sampling Method: Probability Sample
Enrollment: 138 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Hospitalization | baseline
  days
Lymph Nodes number | baseline
  Lymph Nodes number
Clavien Dindo score (post-operative complications) | baseline
  1 to 5 point

SECONDARY OUTCOMES:
Age | Baseline
  years
Body mass index | Baseline
  Kilograms/m2
Lenght of specimen | Baseline
  centimeters

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Gastroenterology IRCCS S. de Bellis, Castellana Grotte, Bari, Italy

IPD SHARING:
Plan to Share IPD: No